CLINICAL TRIAL: NCT01798004
Title: Pilot Study Using Myeloablative Busulfan/Melphalan (BuMel) Consolidation Following Induction Chemotherapy for Patients With Newly Diagnosed High-Risk Neuroblastoma
Brief Title: Busulfan, Melphalan, and Stem Cell Transplant After Chemotherapy in Treating Patients With Newly Diagnosed High-Risk Neuroblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANBL12P1; NCI-2012-02211 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ANBL12P1; COG-ANBL12P1; ANBL12P1 (Other: Children's Oncology Group); ANBL12P1 (Other: CTEP); U10CA180886 (NIH); U10CA098543 (NIH)
Record Dates: First submitted 2013-01-06; First posted 2013-02-25 (Estimated); Results first posted 2017-02-09 (Estimated); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Ganglioneuroblastoma; Stage 1 Neuroblastoma; Stage 2 Neuroblastoma; Stage 2A Neuroblastoma; Stage 2B Neuroblastoma; Stage 3 Neuroblastoma; Stage 4 Neuroblastoma; Stage 4S Neuroblastoma
MeSH Terms: conditions — Ganglioneuroblastoma; Neuroblastoma | interventions — Stem Cell Transplantation; Busulfan; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Cyclophosphamide; Doxorubicin; Etoposide; Congresses as Topic; Radiation; Filgrastim; Granulocyte Colony-Stimulating Factor; Melphalan; Mesna; Peripheral Blood Stem Cell Transplantation; Topotecan; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (induction therapy, consolidation therapy, ASCT) (Experimental): INDUCTION THERAPY:
  COURSES 1-2: Patients receive cyclophosphamide IV over 15-30 minutes and topotecan hydrochloride IV over 30 minutes on days 1-5. Treatment repeats every 3 weeks for 2 courses.
  COURSES 3 AND 5: Patients receive cisplatin IV over 1 hour on days 1-4 and etoposide IV over 1-2 hours on days 1-3. Treatment repeats every 3 weeks for 2 courses.
  COURSE 4: Patients receive cyclophosphamide IV over 1-6 hours on days 1-2, vincristine sulfate IV over 1 minute on days 1-3, and doxorubicin hydrochloride IV over 24 hours on days 1-3. Treatment repeats every 3 weeks for 1 course.
  Treatment continues in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION THERAPY: Beginning 4-8 weeks following the 5th course of induction therapy, patients receive busulfan IV over 3 hours on days -6 to -3 and melphalan IV on day -1. Patients undergo ASCT on day 0.
  Some patients also undergo EBRT after induction and consolidation.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Busulfan; Drug: Cisplatin; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Radiation: External Beam Radiation Therapy; Biological: Filgrastim; Other: Laboratory Biomarker Analysis; Drug: Melphalan; Drug: Mesna; Procedure: Peripheral Blood Stem Cell Transplantation; Other: Pharmacological Study; Drug: Topotecan Hydrochloride; Drug: Vincristine Sulfate

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo autologous peripheral blood stem cell transplant
  Other Names: AHSCT; Autologous; Autologous Hematopoietic Cell Transplantation; Autologous Stem Cell Transplant; Autologous Stem Cell Transplantation; Stem Cell Transplantation, Autologous
Drug: Busulfan — Given IV
  Other Names: 1, 4-Bis[methanesulfonoxy]butane; BUS; Busilvex; Bussulfam; Busulfanum; Busulfex; Busulphan; CB 2041; CB-2041; Glyzophrol; GT 41; GT-41; Joacamine; Methanesulfonic Acid Tetramethylene Ester; Methanesulfonic acid, tetramethylene ester; Mielucin; Misulban; Misulfan; Mitosan; Myeleukon; Myeloleukon; Myelosan; Mylecytan; Myleran; Sulfabutin; Tetramethylene Bis(methanesulfonate); Tetramethylene bis[methanesulfonate]; WR-19508
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
Radiation: External Beam Radiation Therapy — Undergo EBRT
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam Radiotherapy (conventional); External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam; Teleradiotherapy; Teletherapy; Teletherapy Radiation
Biological: Filgrastim — Given SC or IV
  Other Names: Filgrastim Biosimilar Filgrastim-sndz; Filgrastim Biosimilar Tbo-filgrastim; Filgrastim XM02; Filgrastim-aafi; Filgrastim-ayow; Filgrastim-sndz; G-CSF; Granix; Neupogen; Neutroval; Nivestim; Nivestym; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; Releuko; rG-CSF; Tbo-filgrastim; Tevagrastim; XM02; Zarxio
Other: Laboratory Biomarker Analysis — Optional correlative studies
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalan for Injection-Hepatic Delivery System; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
Drug: Mesna — Given IV
  Other Names: 2-Mercaptoethanesulfonate, Sodium Salt; Ausobronc; D-7093; Filesna; Mercaptoethane Sulfonate; Mercaptoethanesulfonate; Mesnex; Mesnil; Mesnum; Mexan; Mistabron; Mistabronco; Mitexan; Mucofluid; Mucolene; UCB 3983; Uromitexan; Ziken
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo autologous peripheral blood stem cell transplant
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood; Peripheral Blood Progenitor Cell Transplantation; PERIPHERAL BLOOD STEM CELL TRANSPLANT; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant; Peripheral Stem Cell Transplantation
Other: Pharmacological Study — Correlative studies
Drug: Topotecan Hydrochloride — Given IV
  Other Names: Evotopin; Hycamptamine; Hycamtin; Nogitecan Hydrochloride; Potactasol; SKF S 104864 A; SKF S-104864-A; SKF S104864A; Topotec; Topotecan HCl; topotecan hydrochloride (oral)
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This pilot clinical trial studies busulfan, melphalan, and stem cell transplant after chemotherapy in treating patients with newly diagnosed neuroblastoma that is likely to come back or spread. Giving chemotherapy to the entire body before a stem cell transplant stops the growth of tumor cells by stopping them from dividing or killing them. After treatment, stem cells are collected from the patient's blood and stored. More chemotherapy or radiation therapy is given to prepare the bone marrow for the stem cell transplant. The stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if the acute toxicity of an autologous stem cell transplant with a busulfan-melphalan (BuMel) based regimen is tolerable when given as consolidation therapy for high-risk neuroblastoma.

EXPLORATORY OBJECTIVES:

I. To determine the incidence of non-hematologic organ toxicity (grade 3 and higher) and all cause mortality in patients undergoing autologous stem cell transplant with a BuMel based regimen followed by local radiotherapy for the treatment of high-risk neuroblastoma.

II. To describe response rates, event-free survival (EFS), and overall survival (OS) for patients undergoing induction therapy followed by consolidation with myeloablative BuMel preparative regimen and local radiotherapy for the treatment of high-risk neuroblastoma.

III. To correlate busulfan pharmacokinetics with non-hematologic toxicity following a BuMel based autologous transplant regimen and event-free survival and overall survival.

IV. To determine the feasibility of performing Curie scores in "real time," as assessed by central scan committee review of a 123 I-meta-iodobenzylguanidine (MIBG) scan obtained after cycle 4 of induction therapy.

V. To examine the concordance between central reviewers and institutional reviewers in performing Curie scoring at diagnosis and after cycle 4 of induction therapy.

VI. To determine the feasibility of detecting aberrations in the anaplastic lymphoma kinase (ALK) gene in tumors obtained at the time of diagnosis in patients with high-risk neuroblastoma.

VII. To determine the feasibility of performing molecular profiling of neuroblastoma tumors obtained at the time of diagnosis in patients with high-risk neuroblastoma.

VIII. To correlate melphalan pharmacokinetics with non-hematologic toxicity following a BuMel based autologous transplant regimen and event-free survival and overall survival.

OUTLINE:

INDUCTION THERAPY:

COURSES 1-2: Patients receive cyclophosphamide intravenously (IV) over 15-30 minutes, topotecan hydrochloride IV over 30 minutes on days 1-5 and filgrastim subcutaneously (SC) or IV once daily (QD) beginning on day 6. Treatment repeats every 3 weeks for 2 courses.

COURSES 3 AND 5: Patients receive cisplatin IV over 1 hour on days 1-4 and etoposide IV over 1-2 hours on days 1-3. Treatment repeats every 3 weeks for 2 courses.

COURSE 4: Patients receive cyclophosphamide IV over 1-6 hours on days 1-2, vincristine sulfate IV over 1 minute on days 1-3, doxorubicin hydrochloride IV over 24 hours on days 1-3 and mesna IV over 15-30 minutes on days 1-2. Treatment repeats every 3 weeks for 1 course.

Treatment continues in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION THERAPY: Beginning 4-8 weeks following the 5th course of induction therapy, patients receive busulfan IV over 3 hours on days -6 to -3 and melphalan IV on day -1. Patients undergo autologous stem cell transplant (ASCT) on day 0 and filgrastim SC or IV beginning on day 0.

Some patients also undergo external beam radiation therapy (EBRT) after induction and consolidation.

After completion of study treatment, patients are followed up every 3 months for 1 year, and then every 6 months for 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of neuroblastoma (International Classification of Diseases for Oncology [ICD-O] morphology 9500/3) or ganglioneuroblastoma (nodular or intermixed) verified by histology or demonstration of clumps of tumor cells in bone marrow with elevated urinary catecholamine metabolites; patients with the following disease stages at diagnosis are eligible, if they meet the other specified criteria
* Patients with newly diagnosed neuroblastoma with International Neuroblastoma Staging System (INSS) stage 4 are eligible with the following:

  * V-myc avian myelocytomatosis viral oncogene neuroblastoma derived homolog (MYCN) amplification (> 4-fold increase in MYCN signals as compared to reference signals), regardless of age or additional biologic features or
  * Age > 18 months (> 547 days) regardless of biologic features or
  * Age 12-18 months (365-547 days) with any of the following 3 unfavorable biologic features (MYCN amplification, unfavorable pathology and/or deoxyribonucleic acid [DNA] index = 1) or any biologic feature that is indeterminate/unsatisfactory/unknown
* Patients with newly diagnosed neuroblastoma with INSS stage 3 are eligible with the following:

  * MYCN amplification (> 4-fold increase in MYCN signals as compared to reference signals), regardless of age or additional biologic features or
  * Age > 18 months (> 547 days) with unfavorable pathology, regardless of MYCN status
* Patients with newly diagnosed neuroblastoma with INSS stage 2A/2B with MYCN amplification (> 4-fold increase in MYCN signals as compared to reference signals), regardless of age or additional biologic features
* Patients with newly diagnosed neuroblastoma with INSS stage 4S with MYCN amplification (> 4-fold increase in MYCN expression signals as compared to reference signals), regardless of additional biologic features
* Patients >= 365 days initially diagnosed with neuroblastoma INSS stage 1, 2, 4S who progressed to a stage 4 without interval chemotherapy; these patients must have been enrolled on ANBL00B1; study enrollment on ANBL12P1 must occur within 4 weeks of progression to stage 4 for INSS stage 1, 2, 4S
* Patients must not have had prior systemic therapy except for localized emergency radiation to sites of life-threatening or function-threatening disease and/or no more than 1 cycle of chemotherapy per a low or intermediate risk neuroblastoma regimen (as per P9641, A3961, ANBL0531, or similar) prior to determination of MYCN amplification status and histology
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * Age 1 month to < 6 months: 0.4 mg/dL
  * Age 6 months to < 1 year: 0.5 mg/dL
  * Age 1 to < 2 years: 0.6 mg/dL
  * Age 2 to < 6 years: 0.8 mg/dL
  * Age 6 to < 10 years: 1 mg/dL
  * Age 10 to < 13 years: 1.2 mg/dL
  * Age 13 to < 16 years: 1.5 mg/dL (males), 1.4 mg/dL (females)
  * Age >= 16 years: 1.7 mg/dL (males), 1.4 mg/dL (females)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age, and
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) or serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) < 10 x ULN for age
* Shortening fraction of >= 27% by echocardiogram, or
* Ejection fraction of >= 50% by radionuclide evaluation
* No known contraindication to peripheral blood stem cell (PBSC) collection; examples of contraindications might be a weight or size less than that determined to be feasible at the collecting institution, or a physical condition that would limit the ability of the child to undergo apheresis catheter placement (if necessary) and/or the apheresis procedure
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Patients that are 12-18 months of age with INSS stage 4 and all 3 favorable biologic features (ie, nonamplified MYCN, favorable pathology, and DNA index > 1) are not eligible
* Female patients who are pregnant are ineligible
* Lactating females are not eligible unless they have agreed not to breastfeed their infants
* Female patients of childbearing potential are not eligible unless a negative pregnancy test result has been obtained
* Sexually active patients of reproductive potential are not eligible unless they have agreed to use an effective contraceptive method for the duration of their study participation

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2013-04-09 (Actual); Primary Completion 2015-07-28 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Meaghan P Granger, Principal Investigator — Children's Oncology Group
Locations (123):
- United States (113):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Maine Children's Cancer Program, Scarborough, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Columbia Regional, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (8):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- Starship Children's Hospital, Grafton, Auckland, New Zealand

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: Induction with multi-agent chemotherapy followed by Consolidation with BuMel chemotherapy + ASCT + XRT
Period: Overall Study
Arm/Group | All Patients
Started | 150
Completed | 63
Not Completed | 87
Not completed — Death | 2
Not completed — Lack of Efficacy | 8
Not completed — Physician Decision | 25
Not completed — Withdrawal by Subject | 4
Not completed — Ineligible | 4
Not completed — Patient/parent refusal | 7
Not completed — Initiation of other non-protocol therapy | 5
Not completed — Enrollment another COG therapeutic trial | 32

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 149
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: Years] | 3.1 [0.4 to 18.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19
  Not Hispanic or Latino | 129
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 21
  White | 107
  More than one race | 0
  Unknown or Not Reported | 11
Region of Enrollment [Number; unit: participants]
  New Zealand | 1
  Canada | 14
  United States | 132
  Australia | 3

OUTCOME MEASURES:

1. Primary Outcome: The Tolerability of BuMel Regimen
Description: Number of patients who experience one or more unacceptable toxicities (severe sinusoidal obstruction syndrome [SOS] or Grade 4-5 pulmonary toxicity per Common Toxicity Criteria [CTC] v.4.0) during the Consolidation phase of therapy.
Time Frame: Up to 28 days post-consolidation therapy, up to 1 year
Population: All eligible and evaluable patients who received at least one dose of either busulfan or melphalan.
Measure: Number; unit: participants
Groups:
- All Patients: Induction with multi-agent chemotherapy followed by Consolidation with BuMel Chemotherapy+ASCT+XRT
Arm/Group | All Patients
Number analyzed (Participants) | 101
participants | 9

2. Other Pre Specified Outcome: Incidence of Non-hematologic Organ Toxicity (Grade 3 and Higher) and All Cause Mortality Graded According to CTC v4.0
Description: Assessed by a descriptive analysis of the incidence of grade 3-5 non-hematologic toxicities (CTC v4.0) and all-cause mortality during consolidation therapy. In addition, a descriptive analysis of "late" onset grade 4-5 pulmonary and hepatic complications that occur within 180 days of the start of consolidation therapy will be examined, regardless if the patient has proceeded to other therapy (including chimeric antibody) during that 180 day period.
Time Frame: Up to 180 days
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Response Rate Determined Using the International Response Criteria
Time Frame: Up to 5 years
Reporting Status: Not Posted

4. Other Pre Specified Outcome: EFS
Time Frame: Up to 5 years
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Overall Survival
Time Frame: Up to 5 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: First Dose Area Under the Curve (AUC) and Average Daily AUC for Busulfan
Description: Relationship with occurrence of non-hematologic toxicities assessed by a descriptive analysis. Association between busulfan exposure levels as measured by the area under the curve (AUC) and event-free survival and overall survival will be examined using Cox proportional hazards models.
Time Frame: Within 28 days following consolidation
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Percentage of Centrally Reviewed Post-course 4 MIBG Scans Reporting a Curie Score Considered to Have Been Determined in "Real Time"
Time Frame: Up to week 12 (course 4 of induction therapy)
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Percentage of MIBG Scans Receiving Institutionally and Centrally Reviewed and Automated Advanced Assisted Scoring Platform Curie Scores Within 1 Unit of Each Other
Description: Cohen's kappa will be calculated to evaluate the concordance in Curie scores between each of the scoring methods at each time point. Up to 160 MIBG scans are expected at diagnosis and up to 144 MIBG scans from the 90% of patients estimated to be MIBG avid are projected post-course 4 of induction therapy, for a total of up to 304 MIBG scans.
Time Frame: Up to week 12 (course 4 of induction therapy)
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Proportion of High-risk Neuroblastoma Patients for Whom ALK Status Can be Obtained
Time Frame: Within 6 weeks of diagnosis
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Proportion of High-risk Neuroblastoma Patients With MYCN Non-amplified Tumors for Whom Molecular Profiling Results Can be Obtained
Time Frame: Within 8 weeks of diagnosis
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Melphalan Pharmacokinetics and the Combination of Busulfan and Melphalan AUC (Optional)
Description: A descriptive analysis of the relationship between melphalan pharmacokinetics and the combination of busulfan and melphalan AUC with the occurrence of non-hematologic toxicities within 28 days following completion of consolidation will be assessed. In addition, the association between melphalan exposure levels as measured by the AUC and event-free survival and overall survival will be examined using Cox proportional hazards models.
Time Frame: Within 28 days post-consolidation
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Four ineligible patients were excluded from the Adverse Event tables, so even though 150 patients enrolled on the study and are summarized in the Participant Flow template, only 146 were at risk for adverse events.
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 10/146
Other Adverse Events (participants affected / at risk) | 82/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=146)
Ascites (Gastrointestinal disorders) | 1 (1)
Death NOS (General disorders) | 2 (2)
Multi-organ failure (General disorders) | 1 (1)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1)
Lung infection (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=146)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 30 (33)
Asystole (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Hearing impaired (Ear and labyrinth disorders) | 5 (6)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Anal pain (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 4 (5)
Colitis (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (5)
Enterocolitis (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (2)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 46 (46)
Nausea (Gastrointestinal disorders) | 8 (9)
Vomiting (Gastrointestinal disorders) | 7 (7)
Fever (General disorders) | 2 (2)
Multi-organ failure (General disorders) | 1 (1)
Pain (General disorders) | 4 (4)
Hepatic pain (Hepatobiliary disorders) | 1 (2)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1)
Portal hypertension (Hepatobiliary disorders) | 2 (2)
Anaphylaxis (Immune system disorders) | 1 (1)
Autoimmune disorder (Immune system disorders) | 1 (1)
Catheter related infection (Infections and infestations) | 4 (6)
Infections and infestations - Other, specify (Infections and infestations) | 11 (13)
Lung infection (Infections and infestations) | 1 (1)
Peritoneal infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 4 (5)
Tracheitis (Infections and infestations) | 1 (1)
Intraoperative arterial injury (Injury, poisoning and procedural complications) | 1 (1)
Intraoperative hemorrhage (Injury, poisoning and procedural complications) | 4 (4)
Intraoperative venous injury (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 7 (8)
Aspartate aminotransferase increased (Investigations) | 9 (10)
Blood bilirubin increased (Investigations) | 13 (15)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
GGT increased (Investigations) | 1 (1)
Investigations - Other, specify (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 4 (5)
Platelet count decreased (Investigations) | 2 (2)
Weight gain (Investigations) | 6 (7)
White blood cell decreased (Investigations) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 28 (34)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (8)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (5)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 27 (35)
Hyponatremia (Metabolism and nutrition disorders) | 5 (5)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (5)
Seizure (Nervous system disorders) | 1 (1)
Vasovagal reaction (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 3 (4)
Thromboembolic event (Vascular disorders) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.